CLINICAL TRIAL: NCT00643864
Title: Mirror-Box Training in Adults With Chronic Hemiparesis Secondary to Stroke: A Descriptive Case Series and Pilot Study
Brief Title: Mirror-Box Training in Adults With Chronic Hemiparesis Secondary to Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-05-14B
Record Dates: First submitted 2008-03-20; First posted 2008-03-26 (Estimated); Results first posted 2019-08-05 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2019-08

CONDITIONS: Stroke
Keywords: mirror training; stroke; hemiparesis; rehabilitation
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mirror training (Other): Training will be performed one-on-one by an investigator in a quiet room, one hour a day, five days a week, for four weeks. The mirror-box apparatus consists of an 18" x 24" vertical mirror secured in the center of a wooden platform. During training, the mirror-box will be placed on a table in front of the subject so that the mirror is perpendicular to the chest, slightly lateral of midline. Subjects will be asked to attend to the mirror reflection of their unaffected hand performing a series of tasks, while keeping their affected limb still. At the end of the four week training period, posttests will be administered by the same therapist who performed the pretests.
  Interventions: Behavioral: mirror training

INTERVENTIONS:
Behavioral: mirror training — Training will be performed one-on-one by an investigator in a quiet room, one hour a day, five days a week, for four weeks. Attendance will be recorded. The mirror-box apparatus consists of an 18" x 24" vertical mirror secured in the center of a wooden platform. During training, the mirror-box will be placed on a table in front of the subject so that the mirror is perpendicular to the chest, slightly lateral of midline. Subjects will be asked to attend to the mirror reflection of their unaffected hand performing a series of tasks, while keeping their affected limb still. At the end of the four week training period, posttests will be administered by the same Occupational Therapist who performed the pretests.

SUMMARY:
The purpose of this project is to assess the effects of four weeks of mirror-box training on weakness of one arm secondary to stroke. Primary measures are function and strength. Secondary measures will evaluate muscle tone, flexibility, and the subject's perception of their everyday function and improvement. Research Hypothesis: For chronic upper limb hemiparesis secondary to stroke, four weeks of mirror-box training with movement of the unaffected limb only results in a mean increase of 10 points on the Fugl-Meyer Test of Motor Recovery (Upper Extremity).

DETAILED DESCRIPTION:
Due to the relatively new nature of mirror training, there are few randomized controlled studies. This pilot case series will serve as our initial step in trying to identify the frequency, duration, and treatment exercises needed in this population. Additionally, this pilot will allow us to ensure our outcome measures are appropriate to detect meaningful treatment changes. After obtaining informed consent, patients will undergo two separate baseline assessments of strength, function, and tone 4 weeks apart. Training sessions will consist of supervised activities using the unaffected arm while observing its mirror reflection; the affected arm will remain still. Sessions will be one hour a day, five days a week, for four weeks. Patients will be tested for strength, function and tone in the affected arm at completion of the four week treatment period by the same occupational therapist that performed the pretests.

ELIGIBILITY:
Inclusion Criteria:

* First unilateral ischemic stroke resulting in hemiparesis at least 6 months prior to enrollment.
* Age at time of enrollment: 30-80 years.
* Voluntary informed consent of patient.
* Patient willing to comply with protocol and is available for all scheduled visits.
* Residual upper extremity hemiparesis.
* No changes in medications planned during 8-week participation.
* No other motor rehabilitative therapy during 8-week participation, including E-stim and acupuncture.
* At least 20 degrees of active wrist extension and 10 degrees of active finger extension against gravity in the affected upper limb, as measured by goniometry.

Exclusion Criteria:

* Serious cognitive deficits, as evidenced by score of <20 on Modified Mini-Mental Status Exam
* Hemorrhagic or bilateral strokes
* Excessive spasticity at the elbow, wrist, or hand, defined as a Modified Ashworth Scale score of >2
* History of botulinum toxin injection in affected upper extremity in the past 4 months
* Lacking >40 degrees of passive elbow extension
* Less than 45 degrees of passive shoulder flexion
* Global or receptive aphasia present on physical exam
* Hemispatial neglect present on physical exam
* Patient participating in constraint-induced therapy during study time period
* Severe visual deficits or visual field deficits as determined by ability to ascertain number of fingers held up on visual field testing
* Deformity/amputation of unaffected upper limb

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2006-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark A Hirsch, PhD, Principal Investigator — CHS; Flora M Hammond, MD, Study Director — CHS
Locations (1):
- Carolinas Rehabilitation, Charlotte, North Carolina, United States

REFERENCES:
- See also: Related Info — http://www.carolinasmedicalcenter.org/body.cfm?id=1571

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Medical outpatient clinic
Groups:
- Mirror Training: Training will be performed one hour a day, five days per week, Monday through Friday, for four weeks.
Period: Pre-test Assessment
Arm/Group | Mirror Training
Started | 3
Completed | 3
Not Completed | 0
Period: Post-test Assessment
Arm/Group | Mirror Training
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Mirror Training: Training will be performed one hour a day, five days a week, Monday through friday, for four weeks.
Arm/Group | Mirror Training
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: The Fugl-Meyer Assessment of Motor Function After Stroke
Description: The Fugl-Meyer Assessment of Motor Function After Stroke, a widely used scale of motor recovery after stroke. The subscale upper extremity motor function was used. This test requires progressively more complex movements and hand grasps and measure speed and coordination. Each item is graded on a 3-point ordinal scale (0=cannot perform; 1=partially performs; 2=performs fully) with a minimum score of 0 and a maximum score of 66 for the upper extremity. Higher scores indicate better outcome.
Time Frame: preintervention and post intervention
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Mirror Training: one group pre post design
Arm/Group | Mirror Training
Number analyzed (Participants) | 3
score on a scale
  Fugl-Meyer Pre | 45.8 (12.6)
  Fugl-Meyer Post | 58 (0)

2. Secondary Outcome: Arm Motor Ability Test
Description: The Arm Motor Ability Test evaluates disabilities in upper extremity function in activities of daily living using a quantitative and qualitative measure. The Functional Ability Scale and the Quality of Movement Scale are rated on an ordinal scale from 0-5. The score for the Functional Ability Scale ranges from 0 to 140. The score for the Quality of Movement Scale ranges from 0 to 140. Higher scores on the Functional Ability and Quality Scale of the Arm Motor Ability Test indicate more normal movement and a better outcome.
Time Frame: preintervention and post intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mirror Training
Number analyzed (Participants) | 3
units on a scale
  Functional Ability Pre | 92.8 (34.8)
  Quality Scale Pre | 90.1 (33.5)
  Functional Ability Post | 98.5 (53.0)
  Quality Scale Post | 94.5 (54.4)

3. Secondary Outcome: Arm Motor Ability Test - Timed
Description: The time in seconds to complete 28 tasks is recorded. The tasks are: 1 pick up utensils, 2 cut meat, 3 fork to mouth, 4 pick up sandwich, 5 sandwich to mouth, 6 pick up spoon, 7 bean in spoon, 8 spoon to mouth, 9 grasp mug handle, 10 mug to mouth, 11pick up comb, 12 comb hair, 13 grasp jar top, 14 open jar, 15 tie lace, 16 phone to ear, 17 press phone number, 18 wipe up water, 19 throw away towel, 20 paretic arm in sleeve, 21 button two buttons, 22 arms in T-shirt, 23 shirt over head, 24 straighten shirt, 25 prop on extended arm, 26 turn on light, 27 open door, 28 close door. The total time in seconds to complete all 28 tasks is recorded - as a total summary score. There is no minimum value. There is no maximum value. Lower scores (e.g., less time to complete the 28 tasks) indicate faster performance and better outcome.
Time Frame: pre intervention and post intervention
Population: One group pre post design
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Mirror Training
Number analyzed (Participants) | 3
seconds
  pre intervention | 330.7 (355.4)
  post intervention | 249.8 (257.2)

ADVERSE EVENTS:
Time Frame: 20 days
Arm/Group | Mirror Training
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes